CLINICAL TRIAL: NCT05781945
Title: COVID-19 Pneumonia and Gut Inflammation: The Role of a Mix of Three Probiotic Strains in Reducing Inflammatory Markers and Need for Oxygen Support
Brief Title: COVID-19 Pneumonia and Gut Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, OJETTI VERONICA, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 3786
Record Dates: First submitted 2023-03-21; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Probiotics; Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic + (Experimental)
  Interventions: Dietary Supplement: probiotics
- standard therapy (Active Comparator)
  Interventions: Other: standard therapy

INTERVENTIONS:
Dietary Supplement: probiotics — supplementation with Bifidobacterium lactis LA 304, Lactobacillus salivarius LA 302,andLactobacillus acidophilus LA 201+ standard theraph for sars-cov-2
  Arms: probiotic +
Other: standard therapy — standard therapy for sars-cov-2
  Arms: standard therapy

SUMMARY:
The primary objective of our study was to evaluate the efficacy of a mix of three probiotic strains (Bifidobacterium lactis LA 304, Lactobacillus salivarius LA 302, and Lactobacillus acidophilus LA 201; Lactibiane Iki®) in the reduction in fecal calprotectin in patients with COVID-19 pneumonia, compared to a control group. The secondary aim was to evaluate the reduction in oxygen support and length of hospital stay in patients taking the probiotic mix.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to our hospital for SARS-CoV-2 infection with respiratory and/or gastrointestinal symptomsandradiological imaging (chest X-ray/CT with/without contrast) of interstitial pneumonia. Patients with mild COVID-19 disease (requiring oxygen support with 2L or 4L nasal cannula or Ventimask 28-35-40% to reach a SpO2-target of 95%)

Exclusion Criteria:

* patients on antibiotic therapy or patients who had taken antibiotics in the previous month; patients with IBD,IBS,or infectious colitis of non-COVID-19 bacterial and/or viral etiology; patients with colonic neoplasia (first to last stage); patients who had undergone colon surgery; patients with severe hepatopathy, nephropathy, heart disease or terminal oncological disease; pregnant women; and patients in circulatory shock and under positive pressure support on admission to hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
efficacy of probiotics in reducing calprotectin and CRP | 10 days
  evaluate the efficacy of a mix of three probiotic strains (Bifidobacterium lactis LA 304, Lactobacillus salivarius LA 302,andLactobacillus acidophilus LA 201) in reducing fecal calprotectin and CRP in patients with COVID-19 pneumonia

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy